CLINICAL TRIAL: NCT06393452
Title: A Randomized, Multicenter, Double-blind, Vehicle-controlled, Phase 2a Study to Assess the Safety, Pharmacokinetics, and Efficacy of PP405 in Adults With Androgenetic Alopecia
Brief Title: Safety, Pharmacokinetics and Efficacy of PP405 in Adults With AGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pelage Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PP405-2001
Record Dates: First submitted 2024-04-26; First posted 2024-05-01 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia | interventions — Gels

STUDY DESIGN:
Intervention Model Description: Subjects who were randomized to vehicle in Part 1 will be eligible to participate in the Open-label Extension in Part 2 of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PP405 0.05% Topical Gel (Active Comparator): 0.05% Topical Gel applied once daily
  Interventions: Drug: PP405 0.05% Topical Gel
- PP405 Topical Vehicle Gel (Placebo Comparator): Placebo Topical Gel applied once daily
  Interventions: Drug: PP405 Topical Vehicle Gel
- PP405 0.05% Topical Gel - Open Label Extension (Other): 0.05% Topical Gel applied once daily for subjects who crossover into the Open-label Extension
  Interventions: Drug: PP405 0.05% Topical Gel

INTERVENTIONS:
Drug: PP405 0.05% Topical Gel — PP405 is an inhibitor of mitochondrial pyruvate carrier (MPC)
  Arms: PP405 0.05% Topical Gel; PP405 0.05% Topical Gel - Open Label Extension
Drug: PP405 Topical Vehicle Gel — PP405 Vehicle = placebo
  Arms: PP405 Topical Vehicle Gel

SUMMARY:
The study is a two part study, designed to validate safety results from the Phase 1 PP405-001 trial while also characterizing longer term safety and PK. Part 1 of the trial is the randomized controlled portion that will focus on safety and PK following 28 days of blinded treatment administration with either PP405 or vehicle control. Part 2 of the trial is an open-label extension that will validate the results of Part 1 with 3 months of treatment administration.

DETAILED DESCRIPTION:
Safety, Pharmacokinetics, and Efficacy Study of PP405 in subjects with Androgenetic Alopecia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 55 years.
2. Able and willing to provide written informed consent.
3. Males must have an AGA modified Norwood-Hamilton Classification score of Type III vertex, Type IV or Type V. Females must have a Savin classification score of I-2, I-3 or I-4.
4. Agree to comply with protocol procedures

Exclusion Criteria:

1. Concomitant diagnosis of non-AGA forms of alopecia.
2. Use of other hair loss treatments within periods specified in protocol.
3. Use of excluded medications as specified in protocol.
4. Diagnosis of other medical conditions as specified in protocol.
5. Any disease or medical condition that, in the opinion of the Investigator, would prevent the subject from participating in the study or might confound study results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-07-16 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-related adverse events | Part 1: Baseline to Day 28; Part 2: Baseline-OLE to Day 84-OLE
  Collection of adverse events, treatment emergent adverse events and serious adverse events.
Change in local dermal tolerability as assessed by subject and investigator | Part 1: Baseline to Day 28; Part 2: Baseline-OLE to Day 84-OLE
  Collection of local skin reactions using a 4 point scale (0-none, 1-mild, 2-moderate, 3-severe)

SECONDARY OUTCOMES:
Pharmacokinetics of PP405 | Part 1: Baseline to Day 28; Part 2: Baseline-OLE to Day 84-OLE
  To assess the concentration of PP405 in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Christina Weng, Study Chair — Pelage Pharmaceuticals
Locations (8):
- United States (8):
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Clinical Trials Research Institute, Thousand Oaks, California
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Minnesota Clinical Study Center, New Brighton, Minnesota
  - DermResearch, Austin, Texas
  - Stride Clinical Research LLC, Sugar Land, Texas
  - Jordan Valley Dermatology Center, South Jordan, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No